CLINICAL TRIAL: NCT05863793
Title: Clinical Study of Acupuncture in the Treatment of Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016LCSY028
Record Dates: First submitted 2023-03-24; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic Peripheral Neuropathy; Acupuncture Treatment
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Acupuncture Group (Experimental): Treatment will be performed by licensed acupuncturists who have at least 5 years of experience in acupuncture. All the acupuncturists will be trained how to locate acupoints, puncture, and manipulate needles before trials.
  Interventions: Other: Acupuncture
- Sham Acupuncture (Sham Comparator): The procedure and duration of treatment in the sham acupuncture group will be identical in the MA group except the needles are blunt tip and there will be no skin penetration and needle manipulation for De qi.
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Other: Acupuncture — The obligatory acupoints include Zhongwan (CV12), bilateral Weiwanxiashu (EX-B3), bilateral Ganshu (BL18), bilateral Pishu (BL20), bilateral Shenshu (BL23), bilateral Zusanli (ST36), bilateral Yanglingquan (GB34), bilateral Sanyinjiao (SP6), bilateral Taixi (KI3), and Bafeng (EX-LE10). Additional acupoints Baxie (EX-UE9) will be added when patients' symptoms appear not only in the lower limbs but also in the upper limbs. After skin disinfection, disposable, stainless steel acupuncture needles will be inserted into the skin of acupoint (approximately 10-20 mm depth), and then manipulations of twirling, lifting, and thrusting will be performed on all needles for at least 10 s to reach De qi (a compositional sensation including soreness, numbness, distention, and heaviness), which is believed to be an essential component for acupuncture efficacy. Needles will be retained in these acupoints for 20 min.
  Arms: Manual Acupuncture Group
Other: Sham Acupuncture — Patients in the SA group will receive sham acupuncture. The procedure and duration of treatment in the SA group will be identical in the MA group except the needles are blunt tip and there will be no skin penetration and needle manipulation for De qi.
  Arms: Sham Acupuncture

SUMMARY:
Diabetic peripheral neuropathy (DPN) is the most common chronic complication of diabetes mellitus that has a considerable impact on quality of life, but there are few effective therapeutic strategies. The aim of this trial is to determine the efficacy and safety of manual acupuncture (MA) versus sham acupuncture (SA) for DPN.

DETAILED DESCRIPTION:
A total of 118 patients with DPN will be recruited and randomly assigned in a 1:1 ratio to either the MA group or SA group. All patients will receive 24 sessions over 12 weeks. Participants will complete the trial by visiting the research center at month 6 for a follow-up assessment. The primary outcome is peroneal motor nerve conduction velocity (peroneal MNCV) at week 12 compared with baseline. Secondary outcomes include peroneal motor nerve action potential amplitude (peroneal MNAP) and latent period (peroneal MNLP), sural sensory nerve conduction velocity (sural SNCV), action potential amplitude (sural SNAP) and latent period (sural SNLP), fasting plasma glucose (FPG), 2-h postprandial blood glucose (2hPG), glycated hemoglobin (HbAlc) at week 12 compared with baseline, Michigan Neuropathy Screening Instrument (MNSI) score and Diabetes Specific Quality of Life scale (DSQL) at week 12 and month 6 compared with baseline. Safety will be assessed during the whole trial. Masking effectiveness will be assessed by patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18-75 years (either sex)
* Patients who meet diagnosis of DPN defined by ADA in 2005：a. DPN is defined as the presence of symptoms and/or signs of peripheral nerve dysfunction in people with diabetes, after the exclusion of other causes. b. NP is defined as altered sensitivity to pressure and (1) altered sensitivity to pain or (2) altered sensitivity to vibration or (3) achilles reflex.
* Symmetric and predominantly sensory, starting from the lower limbs distally and gradually spreading proximally in a glove-and-stocking distribution.
* Ability to understand study procedures and willingness to comply with them for the entire period of study.
* Written informed consent

Exclusion Criteria:

* PN caused by conditions other than diabetes (e.g.,alcohol abuse, chemotherapy, hereditary causes, chronic inflammatory, or idiopathic PN)
* Psychiatric illnesses other than mild depression.
* Severe or unstable cardiovascular, liver, kidney, respiratory, or hematological disorders.
* Received acupuncture treatment in the last 3 months.
* Pregnant or lactating women.
* Research unit personnel directly related to the study and their immediate family members.
* Incapable of giving informed consent or following the study instructions due to language disturbances, serious cognitive deficits, or lack of time.
* Currently participating in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Peroneal Motor Nerve Conduction Velocity | 12 week
  Measurement by electromyography

SECONDARY OUTCOMES:
Glycated hemoglobin (HbA1c) | 12 week
  Observe the changes during the study period
Fasting plasma glucose (FPG) | 12 week
  Observe the changes during the study period
2-h postprandial blood glucose (2hPG) | 12 week
  Observe the changes during the study period
Michigan Neuropathy Screening Instrument (MNSI) score | 12 week
  The MNSI is a clinical and semi-quantitative evaluation of neuropathy that includes medical history and physical assessment. Medical history will be completed by patients with scores ranging between 0 and 13. Physical assessment will be completed by health professionals with five indicators and the aggregate score ranging between 0 and 10: foot appearance (0 and 1 for normal and abnormal, respectively), ulceration (0 and 1 for normal and abnormal, respectively), ankle reflex (0, 0.5, and 1 for normal, reenforced, and absent, respectively), vibration test (0, 0.5, and 1 for normal, weakened, and absent, respectively), and monofilament examination (0, 0.5, and 1 for normal, weakened, and absent, respectively) of feet on both sides.
Quality of life (QoL) | 12 week
  Disease-specific QoL will be assessed at baseline and at week 12, month 6 after randomization using Diabetes Specific Quality of Life scale (DSQL). The scale consists of four domains: interference (12 items), psychology (8 items), social relations (4 items), and treatment (3 items). Each item is measured with a 5-point Likert scale ranging from "not at all" to "extremely". Higher scores indicate worse QoL.
Sural Sensory Nerve Conduction Velocity | 12 week
  Measurement by electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Jian Pei, Study Director — Shanghai University of Traditional Chinese Medicine
Locations (1):
- LongHua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No